CLINICAL TRIAL: NCT00157248
Title: Long-term, Open-label Follow-up Treatment of Patients With Atrial Fibrillation Who Have Been Previously Treated With BIBR 1048 in the PETRO Trial (Trial 1160.20 - NCT01227629). (PETRO Extension Trial: PETRO-Ex)
Brief Title: Long-term, Open-label Follow-up Treatment of Patients With A-fib Who Have Been Previously Treated With BIBR 1048
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Non-Randomized | Masking: None | Purpose: Prevention
Other Study IDs: 1160.42
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2011-02-03 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-02

CONDITIONS: Atrial Fibrillation; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Dabigatran

ARMS (4):
- dabigatran etexilate, 150 mg once daily (Experimental): dosage used at study start
  Interventions: Drug: dabigatran etexilate
- dabigatran etexilate, 150 mg twice daily (Experimental): dosage used at study start
  Interventions: Drug: dabigatran etexilate
- dabigatran etexilate, 300 mg once daily (Experimental): dosage used at study start
  Interventions: Drug: dabigatran etexilate
- dabigatran etexilate, 300 mg twice daily (Experimental): dosage used at study start
  Interventions: Drug: dabigatran etexilate

INTERVENTIONS:
Drug: dabigatran etexilate — dosage used at study start
  Arms: dabigatran etexilate, 150 mg once daily
Drug: dabigatran etexilate — dosage used at study start
  Arms: dabigatran etexilate, 150 mg twice daily
Drug: dabigatran etexilate — dosage used at study start
  Arms: dabigatran etexilate, 300 mg once daily
Drug: dabigatran etexilate — dosage used at study start
  Arms: dabigatran etexilate, 300 mg twice daily

SUMMARY:
To determine the long term safety and efficacy of BIBR 1048 in patients with chronic atrial fibrilla tion, with or without concomitant chronic treatment with acetylsalicylic acid (ASA).

ELIGIBILITY:
Inclusion criteria Diagnosis and main criteria for inclusion: Paroxysmal, persistent, or permanent (chronic) non-rheumatic atrial fibrillation with a history of coronary artery disease (CAD)

Inclusion Criteria:

* previous treatment with BIBR 1048 in PETRO (trial 1160.20- NCT01227629) and no premature discontinuation of therapy
* paroxysmal, persistent, or permanent (chronic) non-rheumatic atrial fibrillation, documented by electrocardiogram (ECG) at least twice prior to enrollment in PETRO
* concomitant coronary artery disease -an additional risk factor for stroke (one or more of the following conditions/events): hypertension, diabetes mellitus (DM), congestive heart failure (CHF) or Left ventricular dysfunction (LVD), previous ischemic stroke or transient ischemic attack) TIA, or age greater than 75 years. -age >= 18 years
* written, informed consent

Exclusion criteria

Exclusion Criteria:

* Valvular heart disease conferring significantly increased risk of thromboembolic events (e.g. clinically significant mitral stenosis or prosthetic valves). planned cardioversion while patients are in the study.
* contraindication to anticoagulant therapy (previous intracranial hemorrhage, gastro-intestinal (GI) hemorrhage within previous 3 months, previous severe hemorrhage with warfarin at therapeutic international normalized ratio (INR), regular use of non-steroidal anti-inflammatory drugs, hemorrhagic diathesis) major bleeding within the last 6 months (other than GI hemorrhage).
* severe renal impairment (estimated glomerular filtration rate [GFR] <= 30 mL/min). uncontrolled hypertension (systolic blood pressure [SBP] > 180 mm Hg and/or diastolic blood pressure [DBP] > 100 mmHg).
* Women who are pregnant or of childbearing potential who refuse to use a medically acceptable form of contraception throughout the study (note: a negative pregnancy test must be obtained for any woman of childbearing potential prior to entry into the study).
* Patients who have received an investigational drug other than BIBR 1048 within the last 30 days.
* Patients considered unreliable by the investigator concerning the requirements for follow-up during the study and/or compliance with study drug administration. Another indication for anticoagulant treatment (eg, deep vein thrombosis or pulmonary embolus). Clinically significant anemia (note: patients with mild-moderate anemia should only be enrolled after the possibility of a GI bleeding source has been evaluated, the etiology of the anemia identified, and appropriate action taken). Patients suffering from thrombocytopenia (platelets < 100,000/uL). Any other condition which, in the discretion of the investigator, would not allow safe participation in the study.
* Continuing or planned concomitant treatment with antiplatelet agents other than acetylsalicylic acid (ASA).
* Recent malignancy or radiation therapy (<= 6 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2003-12; Primary Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (50):
- United States (12):
  - 1160.42.10003 Boehringer Ingelheim Investigational Site, La Mesa, California
  - 1160.42.10006 Boehringer Ingelheim Investigational Site, Pensacola, Florida
  - 1160.42.10004 Boehringer Ingelheim Investigational Site, Port Charlotte, Florida
  - 1160.42.10002 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 1160.42.10015 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1160.42.10008 Boehringer Ingelheim Investigational Site, Westminster, Maryland
  - 1160.42.10012 Boehringer Ingelheim Investigational Site, Pittsfield, Massachusetts
  - 1160.42.10007 Boehringer Ingelheim Investigational Site, Troy, Michigan
  - 1160.42.10014 Boehringer Ingelheim Investigational Site, Hawthorne, New York
  - 1160.42.10013 Boehringer Ingelheim Investigational Site, New Hyde Park, New York
  - 1160.42.10009 Boehringer Ingelheim Investigational Site, North Durham, North Carolina
  - 1160.42.10001 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
- Denmark (13):
  - 1160.42.45010 Boehringer Ingelheim Investigational Site, Aalborg
  - 1160.42.45005 Boehringer Ingelheim Investigational Site, Aarhus C
  - 1160.42.45007 Boehringer Ingelheim Investigational Site, Brædstrup
  - 1160.42.45003 Boehringer Ingelheim Investigational Site, Elsinore
  - 1160.42.45011 Boehringer Ingelheim Investigational Site, Esbjerg
  - 1160.42.45012 Boehringer Ingelheim Investigational Site, Frederikssund
  - 1160.42.45004 Boehringer Ingelheim Investigational Site, Herlev
  - 1160.42.45009 Boehringer Ingelheim Investigational Site, Holbæk
  - 1160.42.45002 Boehringer Ingelheim Investigational Site, Hvidovre
  - 1160.42.45014 Boehringer Ingelheim Investigational Site, Køge
  - 1160.42.45001 Boehringer Ingelheim Investigational Site, Odense
  - 1160.42.45013 Roskilde Sygehus, Roskilde
  - 1160.42.45006 Boehringer Ingelheim Investigational Site, Svendborg
- Netherlands (13):
  - 1160.42.31003 Ziekenhuis Amstelveen, Amstelveen
  - 1160.42.31001 Academisch Medisch Centrum, Amsterdam
  - 1160.42.31013 Onze Lieve Vrouwe Gasthuis, Amsterdam
  - 1160.42.31008 Gelre Ziekenhuis, locatie Juliana, Apeldoorn
  - 1160.42.31006 Wilhelmina Ziekenhuis, Assen
  - 1160.42.31007 Gemini Ziekenhuis, Den Helder
  - 1160.42.31002 Ziekenhuis Gelderse Vallei, Ede
  - 1160.42.31014 Ziekenhuisgroep Twente, Hengelo
  - 1160.42.31012 Vasculair onderzoekscentrum (VOC), Hoorn
  - 1160.42.31009 Havenziekenhuis, Rotterdam
  - 1160.42.31004 Maasland Ziekenhuis, Sittard
  - 1160.42.31005 Tweesteden Ziekenhuis, Tilburg
  - 1160.42.31011 Maxima Medisch Centrum, Veldhoven
- Sweden (12):
  - 1160.42.46013 Boehringer Ingelheim Investigational Site, Eskilstuna
  - 1160.42.46007 Boehringer Ingelheim Investigational Site, Falun
  - 1160.42.46005 Boehringer Ingelheim Investigational Site, Jönköping
  - 1160.42.46010 Boehringer Ingelheim Investigational Site, Kalmar
  - 1160.42.46009 Boehringer Ingelheim Investigational Site, Malmo
  - 1160.42.46008 Boehringer Ingelheim Investigational Site, Norrköping
  - 1160.42.46004 Boehringer Ingelheim Investigational Site, Örebro
  - 1160.42.46002 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.42.46011 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.42.46006 Boehringer Ingelheim Investigational Site, Umeaa
  - 1160.42.46001 Boehringer Ingelheim Investigational Site, Uppsala
  - 1160.42.46003 Boehringer Ingelheim Investigational Site, Västerås

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-randomized open-label extension study of study 1160.20. Patients initially continued Dabigatran treatment of 1160.20; per protocol amendment, most patients moved to 150 mg bid. All events were assigned to the Dabigatran regimen that a patient received prior to the event and patients may be counted in multiple regimens
Pre-assignment Details: In this non-randomized follow-up study, events are displayed cumulatively that occurred in the initial study (1160.20) or in the present study.
Groups:
- Dabigatran Etexilate, 150 mg QD (Once Daily); Dabigatran Etexilate, 150 mg BID (Twice Daily); Dabigatran Etexilate, 300 mg QD (Once Daily); Dabigatran Etexilate, 300 mg BID (Twice Daily): Dosage used at study start
Period: Overall Study
Arm/Group | Dabigatran Etexilate, 150 mg QD (Once Daily) | Dabigatran Etexilate, 150 mg BID (Twice Daily) | Dabigatran Etexilate, 300 mg QD (Once Daily) | Dabigatran Etexilate, 300 mg BID (Twice Daily)
Started | 98 (Started: Participant completed previous trial on Dabigatran and took study drug of present trial.) | 89 | 50 | 124
Completed | 50 (Completed: Participant without premature discontinuation of study medication.) | 52 | 29 | 77
Not Completed | 48 | 37 | 21 | 47
Not completed — Adverse Event | 36 | 25 | 13 | 33
Not completed — Protocol Violation | 4 | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 3 | 3
Not completed — site closures, subject moving | 7 | 7 | 3 | 9

BASELINE CHARACTERISTICS:
Population: All patients in follow-up study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran Etexilate, 150 mg QD (Once Daily) | Dabigatran Etexilate, 150 mg BID (Twice Daily) | Dabigatran Etexilate, 300 mg QD (Once Daily) | Dabigatran Etexilate, 300 mg BID (Twice Daily) | Total
Number analyzed (Participants) | 98 | 89 | 50 | 124 | 361
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.4 (8.6) | 69.3 (8.2) | 71.0 (6.8) | 68.8 (8.5) | 69.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 10 | 12 | 59
  Male | 79 | 71 | 40 | 112 | 302
Atrial fibrillation [Number; unit: Participants] — Atrial fibrillation measured at baseline
  Participants
    Persistent | 40 (139) | 38 (40) | 15 (38) | 46 (15) | 139
    Permanent | 40 | 28 | 25 | 47 | 140
    Paroxysmal | 18 | 23 | 10 | 31 | 82

OUTCOME MEASURES:

1. Primary Outcome: Yearly Event Rate for Composite Endpoint of Stroke, Transient Ischaemic Attacks, System Thromboembolism, Myocardial Infarction, Other Major Adverse Cardiac Events and Mortality.
Description: Time to first occurrence of stroke, transient ischaemic attacks, system thromboembolism, myocardial infarction, other major adverse cardiac events and mortality. Yearly event rate (%) = number of subjects with event / subject-years * 100. Subject years = sum (date of end of treatment - date of start of treatment) of all entered subjects / 365.25
Time Frame: 5 years
Population: All treated patients. In this non-randomized follow-up study, most patients changed treatment regimens per amendment during conduct and treatment exposure was not comparable between regimens. Events were assigned to the regimen a patient received prior to the event, and patients may be counted in multiple regimens. No statistical analysis was done.
Measure: Number; unit: yearly event rate (percentage)
Groups:
- 50 mg Once Daily: Number of Participants treated at any time with 50 mg of Dabigatran etexilate once daily
- 50 mg Twice Daily: Number of Participants treated at any time with 50 mg of Dabigatran etexilate twice daily
- 150 mg Once Daily: Number of Participants treated at any time with 150 mg of Dabigatran etexilate once daily
- 150 mg Twice Daily: Number of Participants treated at any time with 150 mg of Dabigatran etexilate twice daily
- 300 mg Once Daily: Number of Participants treated at any time with 300 mg of Dabigatran etexilate once daily
- 300 mg Twice Daily: Number of Participants treated at any time with 300 mg of Dabigatran etexilate twice daily
Arm/Group | 50 mg Once Daily | 50 mg Twice Daily | 150 mg Once Daily | 150 mg Twice Daily | 300 mg Once Daily | 300 mg Twice Daily
Number analyzed (Participants) | 1 | 105 | 102 | 356 | 90 | 161
yearly event rate (percentage) | 0.0 | 17.0 | 5.0 | 5.7 | 4.5 | 2.4

2. Secondary Outcome: Yearly Event Rate for Stroke
Description: Time to first occurrence of any fatal or non-fatal stroke. Yearly event rate (%) = number of subjects with event / subject-years * 100. Subject years = sum (date of end of treatment - date of start of treatment) of all entered subjects / 365.25
Time Frame: 5 years
Population: as for outcome 1
Measure: Number; unit: yearly event rate (percentage)
Arm/Group | 50 mg Once Daily | 50 mg Twice Daily | 150 mg Once Daily | 150 mg Twice Daily | 300 mg Once Daily | 300 mg Twice Daily
Number analyzed (Participants) | 1 | 105 | 102 | 356 | 90 | 161
yearly event rate (percentage) | 0.0 | 4.3 | 5.0 | 1.1 | 1.7 | 0.0

3. Secondary Outcome: Yearly Event Rate of Ischaemic Stroke
Description: Time to first occurrence of any ischaemic stroke. Yearly event rate (%) = number of subjects with event / subject-years * 100. Subject years = sum (date of end of treatment - date of start of treatment) of all entered subjects / 365.25
Time Frame: 5 years
Population: as for outcome 1
Measure: Number; unit: yearly event rate (percentage)
Arm/Group | 50 mg Once Daily | 50 mg Twice Daily | 150 mg Once Daily | 150 mg Twice Daily | 300 mg Once Daily | 300 mg Twice Daily
Number analyzed (Participants) | 1 | 105 | 102 | 356 | 90 | 161
yearly event rate (percentage) | 0.0 | 4.3 | 5.0 | 0.5 | 1.7 | 0.0

4. Secondary Outcome: Yearly Event Rate of Haemorrhagic Stroke
Description: Time to first occurrence of any haemorrhagic stroke. Yearly event rate (%) = number of subjects with event / subject-years * 100. Subject years = sum (date of end of treatment - date of start of treatment) of all entered subjects / 365.25
Time Frame: 5 years
Population: as for outcome 1
Measure: Number; unit: yearly event rate (percentage)
Arm/Group | 50 mg Once Daily | 50 mg Twice Daily | 150 mg Once Daily | 150 mg Twice Daily | 300 mg Once Daily | 300 mg Twice Daily
Number analyzed (Participants) | 1 | 105 | 102 | 356 | 90 | 161
yearly event rate (percentage) | 0.0 | 0.0 | 0.0 | 0.6 | 0.0 | 0.0

5. Secondary Outcome: Yearly Event Rate for Transient Ischaemic Attacks
Description: Time to first occurrence of any transient ischaemic attacks. Yearly event rate (%) = number of subjects with event / subject-years * 100. Subject years = sum (date of end of treatment - date of start of treatment) of all entered subjects / 365.25
Time Frame: 5 years
Population: as for outcome 1
Measure: Number; unit: yearly event rate (percentage)
Arm/Group | 50 mg Once Daily | 50 mg Twice Daily | 150 mg Once Daily | 150 mg Twice Daily | 300 mg Once Daily | 300 mg Twice Daily
Number analyzed (Participants) | 1 | 105 | 102 | 356 | 90 | 161
yearly event rate (percentage) | 0.0 | 0.0 | 0.0 | 0.2 | 0.4 | 0.0

6. Secondary Outcome: Yearly Event Rate for Systemic Thromboembolism
Description: Time to first occurrence of any non-central nervous system systemic thromboembolism.
  Yearly event rate (%) = number of subjects with event / subject-years * 100. Subject years = sum (date of end of treatment - date of start of treatment) of all entered subjects / 365.25
Time Frame: 5 years
Population: as for outcome 1
Measure: Number; unit: yearly event rate (percentage)
Arm/Group | 50 mg Once Daily | 50 mg Twice Daily | 150 mg Once Daily | 150 mg Twice Daily | 300 mg Once Daily | 300 mg Twice Daily
Number analyzed (Participants) | 1 | 105 | 102 | 356 | 90 | 161
yearly event rate (percentage) | 0.0 | 8.5 | 0.0 | 0.2 | 0.4 | 1.2

7. Secondary Outcome: Yearly Event Rate of Myocardial Infarction
Description: Time to first occurrence of any myocardial infarction. Yearly event rate (%) = number of subjects with event / subject-years * 100. Subject years = sum (date of end of treatment - date of start of treatment) of all entered subjects / 365.25
Time Frame: 5 years
Population: as for outcome 1
Measure: Number; unit: yearly event rate (percentage)
Arm/Group | 50 mg Once Daily | 50 mg Twice Daily | 150 mg Once Daily | 150 mg Twice Daily | 300 mg Once Daily | 300 mg Twice Daily
Number analyzed (Participants) | 1 | 105 | 102 | 356 | 90 | 161
yearly event rate (percentage) | 0.0 | 0.0 | 0.0 | 1.1 | 0.4 | 0.0

8. Secondary Outcome: Yearly Event Rate of Other Major Adverse Cardiac Events
Description: Time to first occurrence of any other major adverse cardiac events. Yearly event rate (%) = number of subjects with event / subject-years * 100. Subject years = sum (date of end of treatment - date of start of treatment) of all entered subjects / 365.25
Time Frame: 5 years
Population: as for outcome 1
Measure: Number; unit: yearly event rate (percentage)
Arm/Group | 50 mg Once Daily | 50 mg Twice Daily | 150 mg Once Daily | 150 mg Twice Daily | 300 mg Once Daily | 300 mg Twice Daily
Number analyzed (Participants) | 1 | 105 | 102 | 356 | 90 | 161
yearly event rate (percentage) | 0.0 | 8.5 | 0.0 | 1.1 | 0.8 | 1.2

9. Secondary Outcome: Yearly Event Rate of Death
Description: Time to death of any cause. Yearly event rate (%) = number of subjects with event / subject-years * 100. Subject years = sum (date of end of treatment - date of start of treatment) of all entered subjects / 365.25
Time Frame: 5 years
Population: as for outcome 1
Measure: Number; unit: yearly event rate (percentage)
Arm/Group | 50 mg Once Daily | 50 mg Twice Daily | 150 mg Once Daily | 150 mg Twice Daily | 300 mg Once Daily | 300 mg Twice Daily
Number analyzed (Participants) | 1 | 105 | 102 | 356 | 90 | 161
yearly event rate (percentage) | 0.0 | 0.0 | 0.0 | 2.7 | 2.1 | 0.0

10. Primary Outcome: Yearly Event Rate for Major Bleeding
Description: Time to first occurrence of fatal or life-threatening, retroperitoneal, intracranial, intraocular, or intraspinal bleeding, which required surgical treatment, led to a transfusion of a minimum of 2 units of packed cells or whole blood, or led to a fall in hemoglobin of 20g/L or less.
  Yearly event rate (%) = number of subjects with event / subject-years * 100. Subject years = sum (date of end of treatment - date of start of treatment) of all entered subjects / 365.25
Time Frame: 5 years
Population: as for outcome 1
Measure: Number; unit: yearly event rate (percentage)
Arm/Group | 50 mg Once Daily | 50 mg Twice Daily | 150 mg Once Daily | 150 mg Twice Daily | 300 mg Once Daily | 300 mg Twice Daily
Number analyzed (Participants) | 1 | 105 | 102 | 356 | 90 | 161
yearly event rate (percentage) | 0.0 | 0.0 | 6.6 | 3.1 | 0.8 | 7.3

11. Primary Outcome: Yearly Event Rate for Major + Minor/Relevant Bleeding
Description: Time to first occurrence of either major or minor/relevant bleeding. Yearly event rate (%) = number of subjects with event / subject-years * 100. Subject years = sum (date of end of treatment - date of start of treatment) of all entered subjects / 365.25
Time Frame: 5 years
Population: as for outcome 1
Measure: Number; unit: yearly event rate (percentage)
Arm/Group | 50 mg Once Daily | 50 mg Twice Daily | 150 mg Once Daily | 150 mg Twice Daily | 300 mg Once Daily | 300 mg Twice Daily
Number analyzed (Participants) | 1 | 105 | 102 | 356 | 90 | 161
yearly event rate (percentage) | 0.0 | 8.5 | 11.6 | 7.6 | 6.6 | 26.8

12. Primary Outcome: Yearly Event Rate for Any Bleeding
Description: Time to first occurrence of any bleeding event. Yearly event rate (%) = number of subjects with event / subject-years * 100. Subject years = sum (date of end of treatment - date of start of treatment) of all entered subjects / 365.25
Time Frame: 5 years
Population: as for outcome 1
Measure: Number; unit: yearly event rate (percentage)
Arm/Group | 50 mg Once Daily | 50 mg Twice Daily | 150 mg Once Daily | 150 mg Twice Daily | 300 mg Once Daily | 300 mg Twice Daily
Number analyzed (Participants) | 1 | 105 | 102 | 356 | 90 | 161
yearly event rate (percentage) | 0.0 | 25.5 | 21.5 | 14.7 | 14.9 | 58.5

13. Secondary Outcome: Yearly Event Rate for Composite Secondary Endpoint of Ischaemic Stroke, Transient Ischaemic Attacks, Non-central Nervous System Systemic Thromboembolism, Myocardial Infarction, Other Major Adverse Cardiac Events and All-cause Mortality
Description: Time to first occurrence of ischaemic stroke, transient ischaemic attacks, non-central nervous system systemic thromboembolism, myocardial infarction, other major adverse cardiac events and all-cause mortality.
  Yearly event rate (%) = number of subjects with event / subject-years * 100. Subject years = sum (date of end of treatment - date of start of treatment) of all entered subjects / 365.25
Time Frame: 5 years
Population: as for outcome 1
Measure: Number; unit: yearly event rate (percentage)
Arm/Group | 50 mg Once Daily | 50 mg Twice Daily | 150 mg Once Daily | 150 mg Twice Daily | 300 mg Once Daily | 300 mg Twice Daily
Number analyzed (Participants) | 1 | 105 | 102 | 356 | 90 | 161
yearly event rate (percentage) | 0.0 | 17.0 | 5.0 | 5.5 | 4.5 | 2.4

14. Secondary Outcome: Severe Adverse Event
Description: Frequency of patients with severe adverse events.
Time Frame: 5 years
Population: All treated patients.
Measure: Number; unit: participants
Arm/Group | 50 mg Once Daily | 50 mg Twice Daily | 150 mg Once Daily | 150 mg Twice Daily | 300 mg Once Daily | 300 mg Twice Daily
Number analyzed (Participants) | 1 | 105 | 102 | 356 | 90 | 161
participants | 0 | 5 | 13 | 96 | 28 | 16

15. Primary Outcome: Yearly Event Rate for Minor Bleeding
Description: Time to first occurrence of minor bleeding. A minor bleeding event is any bleed that does not qualify as a major bleed. All minor bleeding events not fulfilling one of the criteria for clinically relevant were classified as nuisance bleeds.
  Clinically-relevant was defined as spontaneous skin hematoma ≥25 cm², spontaneous nose bleed >5 min, macroscopic hematuria spontaneous or lasting longer than 24 hours if associated with an intervention, spontaneous rectal bleeding, gingival bleeding >5 min, leading to hospitalization, leading to a transfusion of <2 units of packed cells or whole blood and any other bleeding event considered clinically relevant by the investigator.
  Yearly event rate (%) = number of subjects with event / subject-years * 100. Subject years = sum (date of end of treatment - date of start of treatment) of all entered subjects / 365.25
Time Frame: 5 years
Population: as for outcome 1
Measure: Number; unit: yearly event rate (percentage)
Arm/Group | 50 mg Once Daily | 50 mg Twice Daily | 150 mg Once Daily | 150 mg Twice Daily | 300 mg Once Daily | 300 mg Twice Daily
Number analyzed (Participants) | 1 | 105 | 102 | 356 | 90 | 161
yearly event rate (percentage)
  Clinically relevant | 0.0 | 8.5 | 5.0 | 4.5 | 5.8 | 19.5
  Nuisance only | 0.0 | 17.0 | 9.9 | 7.1 | 8.3 | 31.7

16. Secondary Outcome: Laboratory Analyses
Description: Frequency of patients with possible clinically significant abnormalities, i.e. with values out of normal range.
  Normal ranges are defined as:
  * Alanine aminotransferase (ALT): 5-45 [U/L]
  * Aspartate aminotransferase (AST): 10-40 [U/L]
  * Bilirubin, total: 0.2-1.0 [mg/dL]
Time Frame: 5 years
Population: All treated patients.
Measure: Number; unit: participants
Arm/Group | 50 mg Once Daily | 50 mg Twice Daily | 150 mg Once Daily | 150 mg Twice Daily | 300 mg Once Daily | 300 mg Twice Daily
Number analyzed (Participants) | 1 | 105 | 102 | 356 | 90 | 161
participants
  AST > 3*ULN | 0 | 0 | 0 | 10 | 3 | 1
  ALT > 3*ULN | 0 | 0 | 0 | 9 | 4 | 2
  Bilirubin > 2*ULN | 0 | 0 | 0 | 5 | 2 | 0

ADVERSE EVENTS:
Time Frame: 5 years
Description: All treated patients. In this follow-up study, events are displayed cumulatively that occurred in the initial study (1160.20) or in the present study. Most patients changed treatment regimens per amendment during conduct. Events were assigned to the regimen a patient received prior to the event, and patients may be counted in multiple regimens.
Arm/Group | 50 mg Once Daily | 50 mg Twice Daily | 150 mg Once Daily | 150 mg Twice Daily | 300 mg Once Daily | 300 mg Twice Daily
Serious Adverse Events (participants affected / at risk) | 0/1 | 8/105 | 20/102 | 153/356 | 39/90 | 21/161
Other Adverse Events (participants affected / at risk) | 0/1 | 18/105 | 17/102 | 219/356 | 65/90 | 57/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 50 mg Once Daily (N=1) | 50 mg Twice Daily (N=105) | 150 mg Once Daily (N=102) | 150 mg Twice Daily (N=356) | 300 mg Once Daily (N=90) | 300 mg Twice Daily (N=161)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 9 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 1 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 3 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 5 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 6 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 3 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Atrial conduction time prolongation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 12 | 3 | 2
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 6 | 0 | 2
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 3 | 1 | 0
Cardiac asthma (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 2 | 14 | 7 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 2 | 3 | 3 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0
Conduction disorder (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cor pulmonale (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 7 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 3 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 0 | 2 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 3 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 3 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 4 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 7 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 3 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 14 | 1 | 2
Drug ineffective (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysplasia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 3 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 1 | 0
Sudden cardiac death (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 3 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 3 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 2 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0
Gangrene (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Implant site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Meningitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 15 | 2 | 1
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 0 | 0
Implantable defibrillator malfunction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Stent-graft endoleak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure systolic inspiratory decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram ST segment depression (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Heart rate irregular (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 4 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2 | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 3 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 6 | 2 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 3 | 2 | 2 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myasthenic syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 7 | 3 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 3 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Albuminuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Calculus urethral (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal infarct (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urethral haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 0 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 5 | 1 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Prostatism (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 9 | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Joint prosthesis user (Social circumstances) | 0 | 0 | 0 | 1 | 0 | 0
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0
Aneurysm (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0
Aortic aneurysm rupture (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Aortic dissection (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Femoral artery aneurysm (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Femoral artery occlusion (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 4 | 1 | 0
Intermittent claudication (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ischaemia (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Temporal arteritis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Wound haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 50 mg Once Daily (N=1) | 50 mg Twice Daily (N=105) | 150 mg Once Daily (N=102) | 150 mg Twice Daily (N=356) | 300 mg Once Daily (N=90) | 300 mg Twice Daily (N=161)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 21 | 3 | 2
Angina pectoris (Cardiac disorders) | 0 | 1 | 1 | 20 | 8 | 4
Cataract (Eye disorders) | 0 | 0 | 0 | 19 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 1 | 19 | 1 | 4
Constipation (Gastrointestinal disorders) | 0 | 7 | 2 | 14 | 9 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 9 | 4 | 19 | 4 | 6
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 2 | 22 | 3 | 11
Nausea (Gastrointestinal disorders) | 0 | 3 | 2 | 22 | 10 | 6
Chest pain (General disorders) | 0 | 2 | 1 | 18 | 5 | 8
Fatigue (General disorders) | 0 | 2 | 4 | 39 | 12 | 10
Oedema peripheral (General disorders) | 0 | 3 | 6 | 46 | 10 | 8
Bronchitis (Infections and infestations) | 0 | 1 | 2 | 17 | 5 | 3
Influenza (Infections and infestations) | 0 | 1 | 1 | 22 | 9 | 11
Nasopharyngitis (Infections and infestations) | 0 | 3 | 5 | 43 | 13 | 7
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 20 | 3 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 1 | 23 | 3 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 19 | 3 | 11
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 17 | 6 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 5 | 6 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 3 | 2 | 12 | 5 | 6
Gout (Metabolism and nutrition disorders) | 0 | 0 | 3 | 12 | 6 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 6 | 6 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3 | 23 | 6 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 7 | 28 | 13 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 11 | 5 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 5 | 6 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4 | 4 | 18 | 7 | 2
Dizziness (Nervous system disorders) | 0 | 7 | 4 | 36 | 13 | 14
Headache (Nervous system disorders) | 0 | 6 | 3 | 22 | 7 | 5
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 18 | 3 | 2
Haematuria (Renal and urinary disorders) | 0 | 1 | 2 | 32 | 4 | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 6 | 6 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5 | 29 | 15 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 6 | 37 | 12 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 23 | 10 | 11
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 12 | 8 | 3
Haematoma (Vascular disorders) | 0 | 1 | 1 | 17 | 10 | 6
Hypertension (Vascular disorders) | 0 | 2 | 5 | 32 | 14 | 5
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 3 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract